CLINICAL TRIAL: NCT01772056
Title: Randomised Controlled, Double Blind Trial of Topical Twice Weekly Fluticasone Propionate Maintenance Treatment to Reduce Risk of Relapse in Mild or Moderate Atopic Dermatitis in Children
Brief Title: Efficacy Study of Topical Twice Weekly Fluticasone Treatment to Reduce Relapse in Atopic Dermatitis in Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient recruitment is very slow, economic grant has ended and the number of patients is enough according to sample size (22 children/ arm).
Sponsor: Elena Rubio Gomis (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundacion Investigación Hospital General Universitario de Valencia (Unknown)
Responsible Party: Sponsor-Investigator, Elena Rubio Gomis, Professor of Pharmacology. Clinical Pharmacology, University of Valencia
Organization: University of Valencia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FLUTIDANENES08; EC08/00004 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII). Spain); 2008-005360-14 (EudraCT Number)
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, Atopic; Randomized Controlled Trial; Child; Fluticasone; Preventive therapy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone, cream (Experimental): fluticasone propionate (FP) cream of 0.05%. The vehicle is:Base PFCO/W, Propyleneglycol and Water conservant.
  Interventions: Drug: Fluticasone, cream
- Placebo, cream (Placebo Comparator): Vehicle cream is composed by Base PFCO/W, Propyleneglycol and Water conservant.
  Interventions: Drug: Placebo,

INTERVENTIONS:
Drug: Fluticasone, cream — Experimental Group: on treatment with twice weekly on consecutive days FP cream of 0.05% for 16 weeks or at relapse
  Arms: Fluticasone, cream
Drug: Placebo, — Control Group: on treatment with twice weekly on consecutive days vehicle cream for 16 weeks or at relapse.
  Arms: Placebo, cream

SUMMARY:
The relapsing nature of atopic dermatitis (AD) presents a challenge for its long-term treatment. Efficacy and safety of corticosteroids have been proven in the acute treatment of AD, but not its efficacy and security to reduce or prevent relapses.

Objectives To investigate long-term management (16 weeks) of AD with fluticasone propionate (FP) 0,05% cream twice weekly in addition to an emollient (vehicle) after stabilization of an acute flare of AD with FP cream.

DETAILED DESCRIPTION:
Patients 2-10 years of age with a history of mild to moderate AD will be eligible for this multicentre, randomized, double-blind, controlled study if they present an acute flare of AD (<30% affected body surface area; no head). After successful treatment of the flare in an acute phase, patients will receive either, FP twice weekly plus vehicle or vehicle alone over a 16-week maintenance phase. The primary study end point will be probability of a relapse of AD occurring. We will conduct survivor analysis of results.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 2 to 10 years, with mild or moderate acute flare of AD (SCORAD up to 50) and no treatment for this episode of AD.
* written informed consent to patients' parents.

Exclusion Criteria:

* >30% of affected body surface area AD.
* Head affected.
* Fluticasone o vehicle allergy.
* Patients with any medical condition for which topical corticosteroids were contraindicated
* Patients with other dermatological conditions that may have prevented accurate assessment of AD
* Patients with receiving any concomitant medications that might have affected the study's outcome.
* Other medical history that could interfere with the evaluation of study treatment.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Relapse in Atopic Dermatitis (AD). | 16 weeks
  The primary study end point will be probability of a relapse of AD occurring (the relapse rate of AD).

SECONDARY OUTCOMES:
Time to relapse | 16 weeks
  The number of days from start of the Fluticasone propionate treatment in Double-blind Maintenance Phase (DMP) until AD relapse.
Incidence of relapse | 16 weeks
  The proportion of children experiencing a relapse of AD during DMP.
severity of the relapse | 16 weeks
  Severity of AD was scored by means of the modified Scoring of Atopic Dermatitis system (SCORAD).The difference of SCORAD intensity between initial values, Open-label Stabilization Phase (OSP), and end values (end of DMP)
Adverse events and adverse effects | 22 weeks
  Safety was assessed by monitoring adverse events and adverse effects throughout the study.
Therapeutic compliance | 18 weeks
  To describe the therapeutic compliance by means of the control of the drug used.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Rubio Gomis, PhD MD, Principal Investigator — Consorcio Hospital General Universitario de Valencia y Universidad de Valencia
Locations (4):
- Spain (4):
  - Departamento de Salud Valencia-La Ribera, Alzira, Valencia
  - Departamento Valencia-Clinic-Malvarrosa, Valencia, Valencia
  - Departamento de Salud Valencia - Hospital General, Valencia, Valencia
  - Departamento de Salud Valencia-Arnau-Lliria, Valencia, Valencia